CLINICAL TRIAL: NCT01569659
Title: High Dose Lurasidone for Patients With Treatment Resistant Schizophrenia
Acronym: HDL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sunovion Pharmaceuticals
Record Dates: First submitted 2012-03-29; First posted 2012-04-03 (Estimated); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Refractory; Treatment resistant; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose of lurasidone (Active Comparator): Only those patients who still have persistent moderate to severe positive symptoms, even if they have shown some improvement at 80 mg/day will proceed to phase II (randomization). In phase II, 30 subjects will be randomized to continue 80 mg lurasidone.
  Interventions: Drug: Lurasidone
- High dose of lurasidone (Experimental): In phase II, 40 patients will initiate a titration schedule, beginning at 120 mg at week 7. The high-dose group will be increased an additional 40 mg/day every week, thereafter, to a total of 240 mg/day, if adequately tolerated, which would include a worsening of psychopathology as assessed by the PANSS or CGI-S. The dose will remain at 240/day, or the highest dose tolerated, for a duration of 6 months from the time the 120 mg/day dose was initiated.
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — 80 mg/day for up to 30 weeks
  Other Names: Latuda
  Arms: Standard dose of lurasidone
Drug: Lurasidone — Up to 240 mg/day for up to 30 weeks
  Other Names: Latuda
  Arms: High dose of lurasidone

SUMMARY:
The aim of this study is to compare the efficacy of a flexible high dose of lurasidone to a standard dose of lurasidone in patients with treatment resistant schizophrenia or schizoaffective disorder. Efficacy of both dosage groups will be measured through testing of positive symptoms and other components of psychopathology (negative symptoms, general psychopathology, anxiety, depression, cognitive function, global function, severity of illness and tolerability). Patients must qualify for treatment resistance after two or more antipsychotic drug trials to be included in this trial.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a double-blind, randomized trial of lurasidone (80 mg vs 160-240 mg/day) after a 6 week trial of 80 mg/day (phase 1), in treatment resistant adult patients. Only those patients who still have persistent moderate to severe positive symptoms, even if they have shown some improvement at 80 mg/day will proceed to phase II (randomization). In phase II, 30 subjects will be randomized to continue 80 mg lurasidone and 40 will initiate a titration schedule, beginning at 120 mg at week 7. The high-dose group will be increased an additional 40 mg/day every week, thereafter, to a total of 240 mg/day, if adequately tolerated, which would include a worsening of psychopathology as assessed by the PANSS or CGI-S. The dose will remain at 240/day, or the highest dose tolerated, for a duration of 6 months from the time the 120 mg/day dose was initiated. No additional antipsychotic drug of any kind will be permitted in either group during Phase II. Because they are treatment resistant, patients who are doing poorly in either of the two groups in phase II as indicated by level of psychopathology, or as tolerated, and who the clinicians at any site feel should no longer receive lurasidone, will be dropped, and would ordinarily be considered for treatment with clozapine. Where possible, another assessment of these patients, two weeks and four weeks after completion of the trial or early termination will be conducted.

All subjects who enter the phase 1 study will be consented to obtain a blood sample for genetic studies to search for possible markers for response to lurasidone and treatment resistant schizophrenia. DNA from non-treatment resistant patients already studied by the PI will be available for comparison. Following the completion of the study, the PI and the sponsor will discuss how best to analyze the DNA obtained and a separate contract will be written, if indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual IV (DSM-IV) criteria
* All patients must be capable of giving written informed consent.
* The criteria for treatment resistance (TR) will be those of Kane et al, (1988) which are:

  * failure to respond adequately to two or more trials with typical or atypical antipsychotic drugs, of adequate dose and duration (at least 6 weeks) lifetime and at least one such trial within the last two years. No patient with a history of a successful trial of this nature within the last two years will be eligible for inclusion. The minimum doses of antipsychotic drugs permitted in these unsuccessful trials are specified in Table 1.
  * Patients must have scores of 4 (using a 1-7 scale) or more on at least two of the following Positive and Negative Syndrome Scale (PANSS) items: delusions [P1], hallucinations [P3] or unusual thought content [G9]
  * Patients must have a total PANSS score of 70 or above
  * Patients will have had no episodes of good functioning in the previous three years (as defined by current CGI - Severity of moderate to severe, Global Assessment of Functioning (GAF) below 60;
  * Personal and Social Performance Scale of 60 or below.
* Requirement for previous exposure to antipsychotic treatment:

Patients who meet treatment resistance criteria must have had at least two trials with approved antipsychotic drugs, typical or atypical, in the standard dose range. It is recognized that some treatment resistant patients will have had good responses to antipsychotic drugs before meeting treatment resistant criteria.

* All patients must have a Clinical Global Impression - Severity (CGI-S) scale score at screening of at least moderate severity, and must have a Personal and Social Performance (PSP) score of 60 or below.
* Patients may initially be inpatients or outpatients.
* Females of child bearing potential will be admitted only if they are on stable birth control medication and understand that they should not get pregnant during the course of the study. Pregnancy tests will be done at baseline and at approximately 2 month intervals.
* All patients must have stable housing at the current time or will be discharged to a stable outpatient setting for housing, if an inpatient.
* Patients must be willing to remain compliant on oral medication throughout the duration of the trial.

Exclusion Criteria:

* Patients unable to provide written, informed consent
* Patients with a diagnosis other than schizophrenia or schizoaffective disorder.
* Patients currently taking clozapine or have failed an adequate trial of clozapine which lasted at least 2 months.
* Patients who have already failed trials with high doses of other atypical antipsychotic drugs such as risperidone or olanzapine..
* Pregnant females and females who are currently breastfeeding will be excluded.
* Patients with a diagnosis of substance dependence at screening or up to one year prior to enrollment.
* Patients with a history of non-compliance to oral medication to a degree that would interfere with the determination of treatment resistance or diminish likelihood of complying with this protocol
* Patients > age 60
* Uncontrolled medical conditions or recent myocardial infarction or stroke
* BMI =/>45

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2011-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Meltzer, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University Department of Psychiatry and Behavioral Sciences, Chicago, Illinois
  - Northwestern University Psychiatric Clinical Research Program, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karpouzian-Rogers T, Stocks J, Meltzer HY, Reilly JL. The effect of high vs. low dose lurasidone on eye movement biomarkers of prefrontal abilities in treatment-resistant schizophrenia. Schizophr Res. 2020 Jan;215:314-321. doi: 10.1016/j.schres.2019.10.008. Epub 2019 Nov 6. PMID 31706786

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 101 subject were enrolled in phase 1 for a period of 6 weeks to determine Treatment Resistant Status (TRS). 34 determined NOT TRS so were discontinued. The remaining 67 moved to phase 2. 34 remained in standard dose of Lurasidone and 44 were on High dose Lurasidone.
Groups:
- High Dose of Lurasidone: In phase II, 40 patients will initiate a titration schedule, beginning at 120 mg at week 7. The high-dose group will be increased an additional 40 mg/day every week, thereafter, to a total of 240 mg/day, if adequately tolerated, which would include a worsening of psychopathology as assessed by the PANSS or Clinical Global Impressions-Severity (CGI-S). The dose will remain at 240/day, or the highest dose tolerated, for a duration of 6 months from the time the 120 mg/day dose was initiated.
  Lurasidone: Up to 240 mg/day for up to 30 weeks
Period: Overall Study
Arm/Group | Standard Dose of Lurasidone | High Dose of Lurasidone
Started | 34 | 33
Completed | 22 | 22
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose of Lurasidone | High Dose of Lurasidone | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10.7) | 45.2 (11.9) | 46.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive Symptoms of Schizophrenia
Description: Specify Full Scale Name and Construct: Positive and Negative Symptom Scale (PANSS) Scale description: A 45-minute clinical interview is conducted. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers. These 30 items are split into three categories (Positive, Negative and General Psychopathology symptoms of schizophrenia), and the information is used to evaluate the presence, absence and severity of each. A score of 1 on an item indicates the absence of the symptom, up to a 7 which indicates the presence of the symptom is extreme. The minimum and maximum for the whole scale would be 30-210, and for each of the three categories are as follows: Positive scale (7 Items)--minimum score = 7, maximum score = 49; Negative scale (7 Items)--minimum score = 7, maximum score = 49; General Psychopathology scale (16 Items)--minimum score = 16, maximum score = 112.
Time Frame: Baseline to end of randomized phase (24 weeks)
Population: Participants with baseline persistent moderate to severe positive symptoms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Dose of Lurasidone | High Dose of Lurasidone
Number analyzed (Participants) | 34 | 33
units on a scale | 22.6 (3.3) | 24.2 (4.3)

ADVERSE EVENTS:
Arm/Group | Standard Dose of Lurasidone | High Dose of Lurasidone
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/33
Other Adverse Events (participants affected / at risk) | 28/34 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose of Lurasidone (N=34) | High Dose of Lurasidone (N=33)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Fatal cardiac arrest
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose of Lurasidone (N=34) | High Dose of Lurasidone (N=33)
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (9)
Insomnia (Nervous system disorders) | 6 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Suicidality (Nervous system disorders) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Akathasia (Nervous system disorders) | 2 (2) | 3 (3)
Coughing (Infections and infestations) | 2 (2) | 2 (2)
Emesis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Aggression (Nervous system disorders) | 0 (0) | 2 (2)
Hypnatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes